CLINICAL TRIAL: NCT03815435
Title: The Influence of Blood Pressure Upon the Clarity of Surgical Field in Endonasal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KARIM-01-ENSURGERY
Record Dates: First submitted 2019-01-21; First posted 2019-01-24 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
Keywords: Surgical field clarity; Endonasal surgery; Intraoperative bleeding
MeSH Terms: conditions — Disease; Blood Loss, Surgical | interventions — Hypotension, Controlled

STUDY DESIGN:
Intervention Model Description: The study subjects will be enrolled into one arm.
Masking Description: The physician performing the surgery and assessing the surgical field clarity will be masked as to the value of the blood pressure in the individual patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Controlled hypotension (Experimental): Controlled hypotension will be administered according to the clarity of the surgical field evaluated according to the Boezaart scale (1995).
  Interventions: Procedure: Controlled hypotension

INTERVENTIONS:
Procedure: Controlled hypotension — Controlled hypotension will be administered according to the clarity of the surgical field.

SUMMARY:
The work compares the effect of different various values of arterial blood pressure on the clarity of the surgical field in pansinusoperation in patients with chronic rhinosinusitis.

DETAILED DESCRIPTION:
The work compares the effect of different values of arterial pressure on the clarity of the surgical field in pansinus operation in patients with chronic rhinosinusitis. A secondary goal of the study is to compare circulatory parameters, depth of anaesthesia, near-infrared spectroscopy (NIRS) and consumption of hypotensives.

Null hypothesis: There is no difference in the clarity of the surgical field at various levels of the mean arterial pressure.

This study is being realized in accordance with the Declaration of Helsinki and has been approved by the Ethics Committee of the University Hospital Ostrava (849/2018). According to the statement of the State Institute for Drug Control of 26th April 2019 (reference number Sukl96964/2019), the trial is not considered a clinical trial of medicinal products.

Study type: Single-blind study (the surgeon does not know the value of the patient's blood pressure) prospective study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic rhinosinusitis undergoing pansinusoperation
* Age over 18 years
* Concrete surgeon (Petr Matoušek, MD, Ph.D., MBA)
* Concrete anaesthetist (Michal Parma, MD)

Exclusion Criteria:

* Coagulopathy
* Thrombocytopathies
* Vascular wall disorders
* Thrombophlebitis
* Anticoagulation or anti-aggregation therapy
* History of malignancy
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Surgical field clarity in relation to the value of arterial pressure | 13 months
  Clarity of the surgical field will be assessed on a scale of 0-5, according to the Boezaart's system (1995)

SECONDARY OUTCOMES:
Blood pressure | 13 months
  Blood pressure will be measured in the morning before surgery, on arrival at the operating theatre and further 5 minutes after anaesthesia, and every five minutes during the surgery.
Heart rate | 13 months
  Heart rate will be measured in the morning before surgery, on arrival at the operating theatre and further 5 minutes after anaesthesia, and every five minutes during the surgery.
Depth of anaesthesia | 13 months
  Depth of anaesthesia will be measured using the BIS value every 5 minutes
Near infrared spectroscopy (NIRS) | 13 months
  Cerebral perfusion will be measured using the NIRS value every 5 minutes
Consumption of hypotensives | 13 months
  Consumption of hypotensives (Nitro Pohl) will be measured in mg/hr
Blood loss | 13 months
  Blood loss (ml) during the surgery will be measured
Recovery from anaesthesia duration | 13 months
  The interval from the end of surgery to eye opening in minutes will be measured.
Postoperative pain | 13 months
  Postoperative pain will be measured using the VAS (Visual Analogue Scale) upon arrival to the recovery room and the standard ward.
Cognitive function | 13 months
  The standardised clock-drawing test will be performed at the ward, 2 hours after surgery.
Postoperative nausea | 13 months
  The presence of postoperative nausea (YES/NO) will be observed.
Postoperative vomiting | 13 months
  The presence of postoperative vomiting (YES/NO) will be observed.
Complications of controlled hypotension | 13 months
  The presence of complications of controlled hypotension (stroke, myocardial infarction, kidney injury - YES/NO) will be observed.
Use of tamponade | 13 months
  The need to use tamponade due to bleeding (YES/NO) will be observed.
Surgical revision | 13 months
  The need for surgical revision due to bleeding (YES/NO) will be observed.

CONTACTS AND LOCATIONS:
Overall Officials: Ondřej Jor, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Thongrong C, Kasemsiri P, Carrau RL, Bergese SD. Control of bleeding in endoscopic skull base surgery: current concepts to improve hemostasis. ISRN Surg. 2013 Jun 13;2013:191543. doi: 10.1155/2013/191543. Print 2013. PMID 23844295
- [Background] Kelly EA, Gollapudy S, Riess ML, Woehlck HJ, Loehrl TA, Poetker DM. Quality of surgical field during endoscopic sinus surgery: a systematic literature review of the effect of total intravenous compared to inhalational anesthesia. Int Forum Allergy Rhinol. 2013 Jun;3(6):474-81. doi: 10.1002/alr.21125. Epub 2012 Dec 19. PMID 23258603
- [Background] Athanasiadis T, Beule A, Embate J, Steinmeier E, Field J, Wormald PJ. Standardized video-endoscopy and surgical field grading scale for endoscopic sinus surgery: a multi-centre study. Laryngoscope. 2008 Feb;118(2):314-9. doi: 10.1097/MLG.0b013e318157f764. PMID 17989575
- [Background] Milonski J, Zielinska-Blizniewska H, Golusinski W, Urbaniak J, Sobanski R, Olszewski J. Effects of three different types of anaesthesia on perioperative bleeding control in functional endoscopic sinus surgery. Eur Arch Otorhinolaryngol. 2013 Jul;270(7):2045-50. doi: 10.1007/s00405-012-2311-1. Epub 2012 Dec 22. PMID 23263204